CLINICAL TRIAL: NCT01244399
Title: Influence of "Espresso" on Adsorption of Orally Administrated Myo-inositol in Humans
Brief Title: Influence of "Espresso" on Adsorption of Myo-inositol
Status: Completed | Type: Observational
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Collaborators: Azienda istituti Ospitalieri (Unknown)
Other Study IDs: INO_ESP2010
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2011-06

CONDITIONS: Neural Tube Defects
Keywords: inositol; caffeine; NTDs
MeSH Terms: conditions — Neural Tube Defects | interventions — Inositol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

INTERVENTIONS:
Dietary Supplement: Inositol

SUMMARY:
Neural Tube Defects (NTDs) are multifactorial (genetic/environmental) diseases that arise from failure of embryonic neural tube closure. Several studies have demonstrated that periconceptional administration of folic acid can prevent approximately 70% of all NTDs cases. The finding of several NTDs cases in a single family, despite prophylactic therapy with folic acid, suggested that a proportion of human NTDs are folate-resistant. So far, no preventive therapy for folate-resistant NTDs is available. Studies performed on folate-resistant NTDs animal models have shown that inositol is effective in preventing NTDs occurrence. Preliminary results in patients with at least two previous pregnancies affected by NTDs, despite folic acid supplementation, indicate that periconceptional treatment with 500 mg/day of inositol (three months before conception and two months after) is able to prevent NTDs recurrence in humans.

Recently, caffeine intake (more than 10 mg/day) has been associated with an increased risk of NTDs, especially for subgroups of people that carry genetic variants for enzymes involved in caffeine metabolism.

The teratogenic effects of caffeine are known since the 70s. Indeed, gynecologists suggest to pregnant women to avoid/reduce caffeine intake. It is still unknown, however, whether pre-conception caffeine intake interferes with prophylactic therapy for NTDs.

In the proposed study, we aim to evaluate the effect of "espresso" consumption (corresponding to about 100 mg caffeine) on the pharmacokinetics of oral administered myo-inositol (MI), in order to highlight any possible negative effects of caffeine on MI adsorption and excretion before conception.

The study will consist of two phases and will be carried on twelve healthy volunteers. During phase 1, volunteers will be kept for 15 days under inositol-poor diet; at the end of this period, 20 g of MI will be administrated in a single dose. Basal levels of serum and urinary concentration will be evaluated before MI administration (t0); subsequently, sampling will be performed 2, 4, 6 and 8 hours after MI administration. Phase 2 will consist of 15 additional days of inositol-poor diet: basal levels of MI will be again measured before MI administration. In phase 2, MI administration will be concomitant to caffeine exposure through single"espresso" consumption. Samples will be collected at the same time points as in phase 1.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18 to 24

Exclusion Criteria:

* on going pregnancies
* pharmacological treatment in the last 2 weeks
* chronic diseases
* Diabetes

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-11

CONTACTS AND LOCATIONS:
Locations (1):
- Agunco Obstetrics & Gynecology Center, Rome, Italy

REFERENCES:
- [Background] Lorenzo AM, Leon D, Castillo CA, Ruiz MA, Albasanz JL, Martin M. Maternal caffeine intake during gestation and lactation down-regulates adenosine A1 receptor in rat brain from mothers and neonates. J Neurosci Res. 2010 May 1;88(6):1252-61. doi: 10.1002/jnr.22287. PMID 19908252
- [Background] De Castro SC, Leung KY, Savery D, Burren K, Rozen R, Copp AJ, Greene ND. Neural tube defects induced by folate deficiency in mutant curly tail (Grhl3) embryos are associated with alteration in folate one-carbon metabolism but are unlikely to result from diminished methylation. Birth Defects Res A Clin Mol Teratol. 2010 Aug;88(8):612-8. doi: 10.1002/bdra.20690. PMID 20589880
- [Background] Cavalli P, Tedoldi S, Riboli B. Inositol supplementation in pregnancies at risk of apparently folate-resistant NTDs. Birth Defects Res A Clin Mol Teratol. 2008 Jul;82(7):540-2. doi: 10.1002/bdra.20454. No abstract available. PMID 18418886
- [Background] Cavalli P, Copp AJ. Inositol and folate resistant neural tube defects. J Med Genet. 2002 Feb;39(2):E5. doi: 10.1136/jmg.39.2.e5. No abstract available. PMID 11836374
- [Background] van Straaten HW, Copp AJ. Curly tail: a 50-year history of the mouse spina bifida model. Anat Embryol (Berl). 2001 Apr;203(4):225-37. doi: 10.1007/s004290100169. PMID 11396850